CLINICAL TRIAL: NCT06902571
Title: Cross-validating the iTBS-induced Hemodynamic Response From fNIRS and fMRI: a Concurrent iTBS-fMRI-fNIRS Study
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20231218001-03
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy group: A group of healthy adults shall undergo concurrent iTBS/fNIRS/fMRI measurements
  Interventions: Device: Intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta burst stimulation (iTBS) — 600 pulses (3 pulses × 10 bursts × 20 trains = 600 pulses) will be delivered each session with reference to a 3-minute protocol developed by Huang, et al. (2005). Before, during and after iTBS, both fNIRS and fMRI measurements will be conducted simultaneously.

SUMMARY:
Intermittent theta-burst stimulation (iTBS) targeting the left dorsolateral prefrontal cortex (DLPFC) is well established in treating patients with major depressive disorder (MDD). However, the iTBS-induced hemodynamic response during or immediately after a full session of stimulation has not been fully investigated. Although several concurrent iTBS/functional Near Infrared Spectroscopy (fNIRS) and iTBS/functional magnetic resonance imaging (fMRI) studies have investigated the hemodynamic response during or immediately after left DLPFC iTBS, they revealed inconsistent findings in the stimulated DLPFC. Given that the variability in iTBS-induced hemodynamic response in the stimulated DLPFC could be modulated by various inter- and intra-individual factors, cross-validating the findings from both techniques (fNIRS and fMRI) in the same group of participants under the same conditions through a simultaneous fMRI/fNIRS setting enables a straightforward comparison and interpretation of results from each technique. However, to our knowledge, cross-validation of iTBS-related fNIRS and simultaneous fMRI data has not been conducted yet, even the implementation of a simultaneous iTBS/fMRI/fNIRS setup is technically feasible with the mutually compatible equipment. Therefore, the current study has two primary objectives: Firstly, to establish a novel and practical methodological pipeline for simultaneously conducting iTBS/fMRI/fNIRS. Secondly, to cross-validate the hemodynamic responses during and immediately after iTBS, respectively monitored by fNIRS and fMRI.

ELIGIBILITY:
Inclusion Criteria:

* healthiness based on history and psychiatric assessment

Exclusion Criteria:

* a medical history of a major systemic illness or a neurological or psychiatric disorder
* pregnancy
* common fNIRS, MRI and TMS exclusion criteria such as a history of brain surgery, head injury, cardiac pacemaker, intracranial metallic particles or a history of seizures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygenated and deoxygenated hemoglobin (HbO and HbR) change compared to baseline | Before, during and after iTBS stimulation, up to 15 minutes
  iTBS-induced HbO and HbR change in the DLPFC before, during and after stimulation
BOLD signals | Before, during and after iTBS stimulation, up to 15 minutes
  iTBS-induced BOLD change in the DLPFC before, during and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Georg S. Kranz, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No